CLINICAL TRIAL: NCT05387798
Title: A Phase 3, Open-label Extension Study to Assess the Safety, Tolerability, and Efficacy of RAD011 (Cannabidiol Oral Solution) in Patients With Prader-Willi Syndrome
Brief Title: A Phase 3 Extension Study of RAD011 (Cannabidiol Oral Solution) in Patients With Prader-Willi Syndrome
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Program terminated
Sponsor: Radius Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCOUT-016
Record Dates: First submitted 2022-05-17; First posted 2022-05-24 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RAD011 (Experimental)
  Interventions: Drug: RAD011

INTERVENTIONS:
Drug: RAD011 — Cannabidiol Oral Solution (containing synthetic cannabidiol)

SUMMARY:
This is a Phase 3 open-label extension (OLE) study in patients diagnosed with Prader-Willi Syndrome (PWS) who completed the Maintenance Period of the randomized, placebo-controlled Phase 2/3 study SCOUT-015.

The primary objective of this study is to assess the long-term safety and tolerability of RAD011.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a parent/legal guardian that is able to consent for their participation. Parent/caregiver/legal guardian can complete the required assessments throughout the study. Patient Consent/Assent will be obtained if the patient is 8 years of age or older and has the mental capacity to understand and sign a written consent/assent form and/or give verbal assent;
* Patient completed treatment on the SCOUT-015 study through Visit 14 (Week 34);
* If female, is either not of childbearing potential (defined as premenarchal or surgically sterile [bilateral tubal ligation, bilateral oophorectomy, or hysterectomy]) or practicing one of the following medically acceptable methods of birth control up to 4 weeks after the last dose of

RAD011 or placebo:

Exclusion Criteria:

* Significant acute condition (active infection, uncontrolled diabetes, any other uncontrolled chronic condition) including but not limited to clinically significant laboratory abnormality, or medical or psychosocial condition that may preclude the patient from participating in the study, at the Investigator's discretion;
* Positive urine test for drugs of abuse, including tetrahydrocannabinol (THC), or known history of drug, alcohol, or substance abuse;
* Significant risk of committing suicide based on history, psychiatric examination, or based on the Investigator's judgment;
* Significant non-compliance issues (IP misuse or abuse, study visit participation, etc.) during the patient's SCOUT-015 participation based on the Investigator's judgement.
* Pregnant (determined by a positive urine pregnancy test) or lactating female;
* Concurrent participation in any other interventional study involving an investigational product, gene therapy, or device.

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Assess the safety of RAD011 by evaluating the incidence and severity of adverse events reported | Baseline through Week 52
  Safety analyses will be conducted in all subjects who receive at least one dose of RAD011